CLINICAL TRIAL: NCT00987883
Title: Malnutrition and Its Impact on the Perioperational Hospitalization Cost: A Prospective, Cohort Study on Gastroenterological Cancer Patients
Brief Title: The Impact of Perioperational Malnutrition on the Cost on Gastroenterological Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Wei Chen,M.D, Vice Professor, Assisstant Director of Department of Parenteral and Enteral Nutrition, Peking Union Medical College Hospital
Other Study IDs: PUMCH-DPEN-09001
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Malnutrition; Gastroenterological Cancer; Surgical Procedures, Operative
Keywords: Nutritional Support
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Malnutrition cohort: The patients with undernutrition
- Well nourished cohort: Patient that well nourished and without undernutrition

SUMMARY:
Undernutrition is a state marked by energy and/or protein intake deficiency or mal-absorption, and is often described as protein energy malnutrition (PEM). Malnutrition is common in hospitalized patients worldwide. The prevalence of malnutrition in hospitalized patients range from 20% - 50%, depends on the varieties of diseases, health system, population and assessment tools. It is well documented in Western countries that malnutrition affects clinical outcomes negatively. Compared with well-nourished patients, patients with malnutrition stay longer in hospitals and related cost is significantly higher.

There is increasing evidence which indicates that appropriate nutrition support (e.g., standardized nutrition screening procedures, delivering nutrients with appropriate path, etc) may improve clinical outcome on malnutrition, along with cost saving.

To date, there is no study to document specifically the impact of malnutrition and related nutrition support on the health economics in China. Considering China now is on its way to establish public health security system and a diagnosis-related grouping system, the understanding of the cost effectiveness of nutrition support under the current clinical conditions is crucial.

This study aims to investigate the prevalence of perioperational malnutrition in gastroenterological cancer patient, the nutrition support status and related health economic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* With gastroenterological cancer
* Will receive resectional operation
* Consent informed

Exclusion Criteria:

* With severly cardiac, pulmonary, liver or renal disease
* With endocrine or metabolic disease
* With dyslipidemia
* Without consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalization patient in a teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Cost | 30 days after operation

SECONDARY OUTCOMES:
Mortality | 30 days after operation
Infectious morbidity | 30 days after operation
Length of hospitalization | 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, M.D, Study Director — Peking Union Medical College Hospital; Chongmei Lu, M.D, Study Chair — Peking Union Medical College Hospital; Hua Jiang, M.D, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Correia MI, Campos AC; ELAN Cooperative Study. Prevalence of hospital malnutrition in Latin America: the multicenter ELAN study. Nutrition. 2003 Oct;19(10):823-5. doi: 10.1016/s0899-9007(03)00168-0. PMID 14559314
- [Background] Norman K, Pichard C, Lochs H, Pirlich M. Prognostic impact of disease-related malnutrition. Clin Nutr. 2008 Feb;27(1):5-15. doi: 10.1016/j.clnu.2007.10.007. Epub 2007 Dec 3. PMID 18061312
- [Background] Robinson G, Goldstein M, Levine GM. Impact of nutritional status on DRG length of stay. JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):49-51. doi: 10.1177/014860718701100149. PMID 3102782
- [Result] Lochs H, Allison SP, Meier R, Pirlich M, Kondrup J, Schneider S, van den Berghe G, Pichard C. Introductory to the ESPEN Guidelines on Enteral Nutrition: Terminology, definitions and general topics. Clin Nutr. 2006 Apr;25(2):180-6. doi: 10.1016/j.clnu.2006.02.007. Epub 2006 May 11. PMID 16697086